CLINICAL TRIAL: NCT05767892
Title: A Randomized Phase 3 Multicenter Open-Label Study to Compare the Efficacy of YK-029A as First-Line Treatment Versus Platinum-Based Chemotherapy in Patients With Non-Small Cell Lung Cancer With EGFR Exon 20 Insertion Mutations
Brief Title: YK-029A as First-Line Treatment Versus Platinum-Based Chemotherapy for Non-Small Cell Lung Cancer (NSCLC) With EGFR Exon 20 Insertion Mutations
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Puhe Pharmaceutical Technology Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZPH-2023-001
Record Dates: First submitted 2023-03-01; First posted 2023-03-14 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Advanced/Metastatic Non-Small Cell Lung Cancer (NSCLC)
Keywords: NSCLC; EGFR; EXON 20ins
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YK-029A Group (Arm A) (Experimental)
  Interventions: Drug: YK-209A tablet
- Platinum-based Chemotherapy Group (Arm B) (Active Comparator)
  Interventions: Drug: Pemetrexed+carboplatin/Cisplatin

INTERVENTIONS:
Drug: YK-209A tablet — YK-029A 200 milligram (mg) , orally without food，once daily until the participants experience PD as assessed by blinded IRC, intolerable toxicity, or another discontinuation criteria.
  Arms: YK-029A Group (Arm A)
Drug: Pemetrexed+carboplatin/Cisplatin — Participants randomized into chemotherapy arm can receive up to 6 cycles of pemetrexed + carboplatin (pemetrexed 500 mg/m2 + carboplatin area under the plasma concentration-time curve 5 mg/ml per minute (AUC5), IV infusion, every 3 weeks) as the initial treatment. Participants whose disease has not progressed after 4 cycles of first-line platinum-based doublet chemotherapy may receive pemetrexed maintenance monotherapy until a treatment discontinuation criterion is met.
  Arms: Platinum-based Chemotherapy Group (Arm B)

SUMMARY:
The purpose of this study is to compare the effectiveness of YK-029A as first-line treatment with that of platinum-based chemotherapy in participants with locally advanced or metastatic non-small cell lung cancer (NSCLC) whose tumors has epidermal growth factor receptor (EGFR) exon 20 insertion mutations.

Participants will be randomly assigned to one of the two treatment groups YK-029A group or Platinum-based chemotherapy group.

Participants will receive YK-029A orally and pemetrexed/cisplatin or pemetrexed/carboplatin via vein until the participants experience worsening disease (PD) as assessed by blinded independent review committee (IRC), intolerable harmful effects or another discontinuation criteria.

DETAILED DESCRIPTION:
The drug being tested in this study is called YK-029A. YK-029A is being tested to evaluate the efficacy as a first line treatment compare with platinum-based chemotherapy in the participants with locally advanced or NSCLC whose tumors harbor EGFR exon 20 insertion mutations.

The study will enroll 350 patients. Participants will be randomly assigned to one of the two treatment groups-YK-029A Group (Arm A) or Platinum-based Chemotherapy Group (Arm B).

The participants will be administered with YK-029A orally in arm A and pemetrexed/cisplatin or pemetrexed/carboplatin intravenously (IV) in arm B until the participants experience progressive disease (PD) as assessed by blinded independent review committee (IRC), intolerable toxicity or another discontinuation criteria.

Participants in the chemotherapy group should not be allowed to cross over to treatment with YK-029A after IRC-assessed PD is documented. Randomized treatment with YK-029A or platinum-based chemotherapy may be continued after PD, at the discretion of the investigator and with the sponsor's approval, if there is still evidence of clinical benefit.

This multi-center trial will be conducted in China . The overall time to participate in this study is until 3 years after the last participant is randomized. Participants will make multiple visits to the clinic and will be followed for survival, subsequent anticancer therapy, subsequent disease assessment outcome until disease progression on a subsequent anticancer therapy, and participant-reported health status (EORTC QLQ-C30 and EORTC QLQ-LC13) for 3 years after the last participant is randomized in the study and 30 days after the last dose of study drug for safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult patients (aged 18 years or older).
2. Histologically or cytologically confirmed nonsquamous cell locally advanced not suitable for definitive therapy, recurrent, or metastatic (Stage IV) NSCLC.
3. Documented epidermal growth factor receptor (EGFR) in-frame exon 20 insertion mutation assessed by a clinical laboratory improvements amendment (CLIA)-certified (China sites) or an accredited (outside of the US) local laboratory.

3、The EGFR exon 20 insertion mutation can be either alone or in combination with other EGFR or human epidermal growth factor receptor 2 (HER2) mutations except EGFR mutations for which there are approved anti-EGFR tyrosine kinase inhibitors [TKIs] (ie, exon 19 del, L858R, T790M, L861Q, G719X, or S768I, where X is any other amino acid).

4、Adequate tumor tissue available, either from primary or metastatic sites, for central laboratory confirmation of EGFR exon 20 insertion mutation.

5、At least 1 measurable lesion per RECIST Version 1.1. 6、Life expectancy ≥3 months. 7、Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. 8、Adequate organ and hematologic function as defined by blood transfusions with a recommended >/ 14 day washout period.

Exclusion Criteria:

1. Received prior systemic treatment for locally advanced or metastatic disease, including local administration, such as intra-pleural injection of anticancer medication with the exception noted below.
2. Neoadjuvant or adjuvant chemotherapy/immune therapy for Stage I to III or combined modality chemotherapy/radiation for locally advanced disease is allowed if completed >6 months before the development of metastatic disease.
3. Received radiotherapy ≤14 days before randomization or has not recovered from radiotherapy-related toxicities.
4. Received a moderate or strong cytochrome P450 (CYP)3A inhibitor or moderate or strong CYP3A inducer within 10 days before first dose of YK-029A.
5. Concurrent EGFR mutations: exon 19 deletion, L858R, T790M, G719X, S768I, or L861Q.
6. Have been diagnosed with another primary malignancy other than NSCLC。
7. Have current spinal cord compression or leptomeningeal disease.
8. Have uncontrolled hypertension. Participants with hypertension should be under treatment on study entry to control blood pressure.
9. Received a live vaccine within 4 weeks before randomization per Summary of product characteristics (SmPCs) for pemetrexed, cisplatin, and carboplatin.
10. As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses (i.e., hemophilia and Von Willebrand disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18 Years and older (Adult, Older Adult)
Enrollment: 350 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) as Assessed by Blinded Independent Review Committee (IRC) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 . | Up to approximately 36 months after the first participant is randomized.
  PFS is defined as the time interval from the date of randomization until the first date at which the criteria for progressive disease (PD) according to RECIST Version 1.1 are met or death, whichever occurs first.

SECONDARY OUTCOMES:
Confirmed Objective Response Rate (ORR) as Assessed by Blinded Independent Review Committee (IRC) per RECIST Version 1.1 | Up to approximately 36 months after the first participant is randomized.
  Confirmed ORR is defined as the percentage of participants who are confirmed to have achieved complete response (CR) or partial response (PR). Confirmed responses are responses that persist on repeat imaging ≥4 weeks after initial response.
Overall Survival (OS) | Up to approximately 36 months after the first participant is randomized.
  OS is defined as the interval from the date of randomization until death.
Progression Free Survival (PFS) as Assessed by the Investigator | Up to approximately 36 months after the first participant is randomized.
  PFS is defined as the time interval from the date of randomization until the first date at which the criteria for PD according to RECIST Version 1.1 are met or death, whichever occurs first.
Confirmed Objective Response Rate (ORR) as Assessed by the Investigator | Up to approximately 36 months after the first participant is randomized.
  Confirmed ORR is defined as the percentage of participants who are confirmed to have achieved CR or PR. Confirmed responses are responses that persist on repeat imaging ≥4 weeks after initial response.
Duration of Response, as Assessed by the Blinded Independent Review Committee (IRC) and the Investigator. | Up to approximately 36 months after the first participant is randomized.
  Duration of response is defined as the time interval from the time that the measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that PD or death (whichever occurs first) is objectively documented.
Disease Control Rate (DCR) as Assessed by the Blinded Independent Review Committee (IRC) and the Investigator | Up to approximately 36 months after the first participant is randomized.
  DCR is defined as the percentage of participants who have achieved CR, PR, or stable disease (SD) (in the case of SD, measurements must have met the SD criteria at least once after study entry at a minimum interval of 6 weeks) after the initiation of study drug.
Patient-reported Symptoms, Functioning, and Health-related Quality of Life (HRQoL) as Assessed by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 | Up to approximately 36 months after the first participant is randomized.
  EORTC QLQ-C30 is a cancer-specific questionnaire which comprises of 5 functional scales (physical, role, cognitive, emotional, and social functioning); 3 symptom scales (fatigue, pain, and nausea/vomiting); and a global health status/quality-of-life (QoL) scale. Six single-item scales are also included (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Raw scores will be converted into scale scores ranging from 0 to 100. For the functional scales and the global health status/QoL scale, higher scores represent better HRQoL, whereas for the symptom scales lower scores represent better HRQoL (i.e., a low level of symptomatology/problems).
Participant-reported Symptoms as Assessed by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire, Lung Cancer Module (QLQ-LC13). | Up to approximately 36 months after the first participant is randomized.
  EORTC QLQ-LC13 is a cancer-specific questionnaire which comprises of 13 questions assessing lung cancer-associated symptoms (cough, hemoptysis, dyspnea, and site-specific pain), treatment-related side effects (sore mouth, dysphagia, peripheral neuropathy, and alopecia), and use of pain medication. Raw scores will be converted into scale scores ranging from 0 to 100. Higher scores represent a high level of symptomatology/problems.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zhao, Doctor, Study Director — Puhe Biopharma
Locations (52):
- China (52):
  - The First Affiliated Hospital of Bengbu Medical Colleg, Bengbu, Anhui
  - Anhui Provincial Chest Hospital, Hefei, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - Yijishan Hospital of Wannan Medical College, Wuhu, Anhui
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Cancer Hospital Affiliated to Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - People's Hospital of Zhongshan City, Zhongshan, Guangdong
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - he First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhenzhou, Henan
  - Tongji Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Third Xiangya Hospital, Central South University, Changsha, Hunan
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow Universit, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Jilin Provincial Cancer Hospital, Changchun, Jilin
  - he First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Cancer Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - the First Affiliated Hospital; Medical College of Xi'an Jiaotong University, Xian, Shanxi
  - The Second Affiliated Hospital of PLA Air Force Medical University, Xian, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Cancer in Zhejiang Province, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Taizhou First People's Hospital, Taizhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - Peking Union Medical College Hospital, Beijing
  - National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing
  - Peking University Cancer Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No